CLINICAL TRIAL: NCT03096535
Title: Cold Induced Activation of Brown Fat in Humans Assessed With PET/MR Scans and Skin-temperature Measure - A Cross-over Randomized Controlled Trial.
Brief Title: Cold Induced Activation of Brown Adipose Tissue in Humans
Acronym: COLDBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susanna Søberg (Other)
Responsible Party: Sponsor-Investigator, Susanna Søberg, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-16038581-COLDBAT
Record Dates: First submitted 2017-02-23; First posted 2017-03-30 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Adipose Tissue, Brown; Brown Adipose Tissue; Brown Fat; Uncoupling Protein 1; Adipokines; Proteomics; Infrared Thermography; BAT; Obesity; Type 2 Diabetes; Proteins
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Cool-Down Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooling (Experimental): Individualized cooling protocol.
  Interventions: Procedure: Cooling
- Thermoneutral (Experimental): Thermoneutral condition day.
  Interventions: Procedure: Thermoneutral

INTERVENTIONS:
Procedure: Cooling — Individualized cooling protocol.
  Other Names: Cold activation; Cold stimulation; Cold activation of BAT
  Arms: Cooling
Procedure: Thermoneutral — Thermoneutral control day.
  Arms: Thermoneutral

SUMMARY:
This study investigates cold-induced brown fat activation assessed using PET/MR scans. Subjects will participate in an acute cooling intervention day and a thermoneutral intervention day with PET/MR scans on both days. A secondary purpose is to make a validation of an infrared thermography camera by comparison of skin temperatures and SUV of the supraclavicular brown adipose tissue.

DETAILED DESCRIPTION:
The field of human brown adipose tissue (BAT) research is focused on activation of BAT as a means of manipulating energy expenditure and potentially anti-obesity and anti-diabetic properties of the tissue. This is well established in rodent studies and explained as due to the specific brown fat uncoupling protein 1 (UCP1). Despite increasing evidence that indicates a metabolic regulatory role of BAT in humans, BAT activation/recruitment is not fully understood and even less is known about the endocrine capacities of human BAT.

Cold induced brown fat activity will be assessed with PET/MR scans and validate an infra-red thermography camera, as well as perform a proteomic screening using blood samples under these two intervention days.

15 healthy lean male subjects will serve as their own control in a cross-over randomized control study, including a pre-examination day, a thermoneutral-day and a cooling test-day with cold exposure followed by a PET/MR scan to determine BAT activity. An extra cooling day is applied for the external validation of the infrared thermography camera. Blood samples and abdominal fat-biopsies will be taken at thermoneutral condition and under cold stimulation of brown fat.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-30 years.
* Men
* Caucasian white
* Body Mass Index 19-25 kg/m2.
* Moderate physical activity level (not more than 8-10 hours of training pr. Week)
* Ability to give informed consent.
* Ability to follow verbal and written instructions in Danish.
* Body fat percent under 21% measured at the pre-examination day.

Exclusion Criteria:

* Chronic diseases: Hormonal: Metabolic Diseases mb. Graves, hypothyroidism, myxedema and goiter. Diabetes Melitus, Coronary heart disease (history of myocardial infarction, unstable angina pectoris, or congestive heart failure), cancer treated within last 3 years.
* Tobacco, marijuana or intravenous drug use within 1 year of screening.
* Dieting, recent weight loss (>3 kg within 3 month) or a history of an eating disorder.
* Dietary supplements.
* History of depression, psychosis, or other psychiatric illness requiring hospitalization.
* Alcohol consumption >14 units/week.
* History of alcohol abuse within the past 3 years.
* Known liver disease or elevated liver biomarkers more than 2 times upper normal levels in the preliminary investigation.
* Known kidney disease or elevated kidney biomarkers, eCRF <60 ml/min, in the preliminary investigation.
* Use of daily medications, except for seasonal use of antihistamines.
* Diagnosed sleep disturbances.
* Pacemaker or other electronics implanted in the body.
* Magnetic impressionable metal implants or foreign objects in the body inconsistent with completion of MR.
* Claustrophobia
* Communication problems, including understanding the experimental protocol
* History of contrast allergy.
* Winter swimmers.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-02 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Difference in brown adipose tissue (BAT) activity after cooling versus no cooling. | Difference in SUV mean after 2 hours of cooling versus 2 hours of no cooling.
  BAT activity is measured by standard fluorodeoxyglukose uptake volume (SUV mean) in the supraclavicular BAT depot using PET/MR scans. Difference between scans performed after 2 hours of cooling and 2 hours of no cooling is calculated.

SECONDARY OUTCOMES:
Difference in BAT activity after cooling versus no cooling. | Difference in peak temperature after 2 hours of cooling versus 2 hours of no cooling.
  BAT activity is measured by skin temperature in the supraclavicular BAT depot using infrared thermography imaging. Difference between peak temperature change (peak temperature minus baseline temperature) during 2 hours of cooling and 2 hours of no cooling is calculated.
Difference in resting energy expenditure after cooling versus no cooling | Difference in resting energy expenditure after 2 hours of cooling versus 2 hours of no cooling.
  Difference in resting energy expenditure after cooling versus no cooling, measured as mean difference in KJ/min.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Søberg, MSc., Principal Investigator — Center for Inflammation and Metabolism/Center for physical activity research
Locations (1):
- Center for Inflammation and Metabolism/ Center for Physical Activity Research, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soberg S, Lofgren J, Philipsen FE, Jensen M, Hansen AE, Ahrens E, Nystrup KB, Nielsen RD, Solling C, Wedell-Neergaard AS, Berntsen M, Loft A, Kjaer A, Gerhart-Hines Z, Johannesen HH, Pedersen BK, Karstoft K, Scheele C. Altered brown fat thermoregulation and enhanced cold-induced thermogenesis in young, healthy, winter-swimming men. Cell Rep Med. 2021 Oct 11;2(10):100408. doi: 10.1016/j.xcrm.2021.100408. eCollection 2021 Oct 19. PMID 34755128